CLINICAL TRIAL: NCT00848302
Title: Endothelial Function in Human Arteries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23HLOBO247; K23HLOBO247 (Other: National Heart Lung Blood Institute)
Record Dates: First submitted 2009-02-12; First posted 2009-02-20 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Endothelial Dysfunction
Keywords: peripheral vascular disease; endothelial dysfunction; intravascular ultrasound; L-Arginine
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Arginine; Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-arginine (Experimental): Assess the effects of regional L-arginine supplementation in patients with chronic lower extremity occlusive disease undergoing angiography
  Interventions: Drug: L-arginine

INTERVENTIONS:
Drug: L-arginine — 30 patients will receive either 50, 100 or 500mg L-arginine supplementation infused via a end-hole catheter
  Other Names: Nitric oxide

SUMMARY:
Up to 30 patients with lower extremity disease scheduled to undergo diagnostic angiography will undergo baseline bloodwork and IVUS (intravascular ultrasound), followed by dosing with L-arginine to assess changes in endothelial function.

DETAILED DESCRIPTION:
We will assess doses of regional L-arginine supplementation in patients undergoing elective angiography for lower extremity PAD. Assessment of EDR and EIR with IVUS in patent arteries will be performed with one of 3 doses of catheter-directed L-arginine. We will obtain plasma samples from the peripheral arteries and assay amino acid levels and protein oxidation products using mass spectrometry. These experiments will determine the optimal L-arginine supplementation dose to be used in further studies. We expect to show that L-arginine supplementation will have a more significant effect on vessels less affected by atherosclerosis, but that this effect diminishes with greater atheroma accumulation as measured by IVUS virtual histology. Also, we expect L-arginine supplementation to be most effective in vessels with low baseline L-arginine levels. Lastly, we will compare local arterial factors obtained via catheter-directed arterial sampling (NOx, L-arginine, nitrotyrosine levels) to traditional serum risk factors (glucose, HbA1c, LDL, homocysteine and hs C-reactive protein).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* symptoms of intermittent claudication, rest pain or minor tissue loss (Rutherford Category I-V)
* ABI of <.90
* angiographic demonstration of a 100mm patent segment of superficial femoral artery containing at least one distal runoff vessel

Exclusion Criteria:

* acute limb ischemia,
* contraindication to angiography (creatinine >2.5)
* concurrent oral anticoagulant therapy that cannot be safely withheld
* extensive tissue loss or gangrene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
IVUS mediated assessment of endothelial-dependent (EDR) and endothelial-independent (EIR) vasorelaxation before and after catheter-directed L-arginine delivery in patent arteries. | Procedural

SECONDARY OUTCOMES:
Local arterial factors including peripheral L-arginine and nitrotyrosine levels via mass spectrometry and morphologic parameters of plaque composition. | Procedural

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Kashyap, MD, Principal Investigator — Cleveland Clinic Vascular Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kashyap VS, Lakin RO, Campos P, Allemang M, Kim A, Sarac TP, Hausladen A, Stamler JS. The LargPAD Trial: Phase IIA evaluation of l-arginine infusion in patients with peripheral arterial disease. J Vasc Surg. 2017 Jul;66(1):187-194. doi: 10.1016/j.jvs.2016.12.127. Epub 2017 Mar 30. PMID 28366306
- [Derived] Kashyap VS, Lakin RO, Feiten LE, Bishop PD, Sarac TP. In vivo assessment of endothelial function in human lower extremity arteries. J Vasc Surg. 2013 Nov;58(5):1259-66. doi: 10.1016/j.jvs.2013.05.029. Epub 2013 Jul 3. PMID 23830159